CLINICAL TRIAL: NCT01273792
Title: Investigation of Relevant Biomarkers in Patients With Susac Syndrome
Brief Title: Investigation of Biomarkers in Susac Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jan-Markus Dörr, PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: Biomarkers Susac Syndrome
Record Dates: First submitted 2011-01-06; First posted 2011-01-11 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Susac Syndrome
MeSH Terms: conditions — Susac Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (serum, Blood cells)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Susac syndrome
- Matched healthy controls

SUMMARY:
Susac Syndrome is a rare disease and the establishment of the diagnosis is often difficult. The aim of this investigation is to identify relevant biomarkers and to elucidate the pathogenesis of Susac syndrome

DETAILED DESCRIPTION:
Susac Syndrome is a rare disease characterized by encephalopathy, branch retinal artery occlusion and sensorineural deafness. The pathogenesis is not yet clear, an autoimmune endotheliopathy is discussed. Because of the variable and often incomplete clinical presentation, the establishment of the diagnosis is often delayed or even completely missed.

The aim of this study is to identify biomarkers that facilitate the reliable and prompt establishment of the diagnosis. Patients with a definite diagnosis of Susac syndrome and healthy subjects as controls are investigated.

Furthermore, the correlation of serological markers with structural retinal and cerebral changes will contribute to clarification of the pathogenesis of Susac syndrome.

ELIGIBILITY:
Inclusion Criteria:

* adult male and female patients with definite Susac syndrome or matching healthy control subjects
* ability to provide informed consent

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with Susac syndrome (male/female; healthy control subjects
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
disease specific patterns of pathology on cranial MRI
  one-time cranial MRI
disease specific patterns of pathology in optical coherence tomography
  one time optical coherence tomography
serological biomarkers | not defined, cross-sectional analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Dörr, MD, Principal Investigator — NeuroCure Clinical Research Center, Charité Universitaetsmedizin Berlin
Locations (1):
- NeuroCure Clinical Reserach Center, Charité Universitaetsmedizin, Berlin, Germany

REFERENCES:
- [Background] Dorr J, Radbruch H, Bock M, Wuerfel J, Bruggemann A, Wandinger KP, Zeise D, Pfueller CF, Zipp F, Paul F. Encephalopathy, visual disturbance and hearing loss-recognizing the symptoms of Susac syndrome. Nat Rev Neurol. 2009 Dec;5(12):683-8. doi: 10.1038/nrneurol.2009.176. PMID 19953118